CLINICAL TRIAL: NCT02752061
Title: Potlako: A Programmatic Multi-facility Level Intervention to Improve Access to Timely Oncology Care in Botswana
Brief Title: Potlako: A Programmatic Intervention to Improve Access to Timely Oncology Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Brigham and Women's Hospital (Other); Botswana Harvard AIDS Institute Partnership (Other); Botswana Ministry of Health (Other Government); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Scott Dryden-Peterson, Assistant Professor, Research Affiliate, Harvard School of Public Health (HSPH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BHP078
Record Dates: First submitted 2016-04-22; First posted 2016-04-26 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Neoplasms; HIV; Healthcare Disparity
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kweneng East District (Experimental): Patient presenting with possible cancer symptoms/sign to a clinic or hospital in Kweneng East District during study period.
  Interventions: Other: Potlako intervention
- All other districts (No Intervention): Patient presenting with possible cancer symptoms/sign to a clinic or hospital in all other districts of Botswana (or Kweneng East prior to implementation of intervention).

INTERVENTIONS:
Other: Potlako intervention — Multicomponent intervention including:
  * provider training on early detection and diagnostic approaches to cancer
  * patient education on importance of obtaining timely cancer diagnosis
  * provision of a patient navigator to facilitate diagnosis and entry into care
  * provision of transportation support to vulnerable patients
  Arms: Kweneng East District

SUMMARY:
Diagnostic and treatment delays contribute substantially to disparities in cancer morbidity and mortality between low- and middle- income countries (LMICs) and high-income countries. Individuals present with advanced stage disease resulting in minimal chance for cure or long-term survival.

The Potlako project will implement and evaluate a multifaceted intervention to test the hypothesis that a package of enhanced coordination of care including an electronic messaging, transportation support, and training targeted at generalist clinicians at primary and secondary level facilities, can reduce time to diagnosis and stage at diagnosis for HIV-infected individuals with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Citizen of Botswana
* Suspected or diagnosed cancer

Exclusion Criteria:

* Involuntary incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 979 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Cancer stage | 1 day visit
Time from initial clinic visit with cancer symptom/sign to entry into oncology care | 1 day visit

CONTACTS AND LOCATIONS:
Locations (1):
- Botswana Harvard AIDS Institute, Gaborone, Botswana

REFERENCES:
- [Derived] Tapela NM, Peluso MJ, Kohler RE, Setlhako II, Botebele K, Gabegwe K, Nkele I, Narasimhamurthy M, Mmalane M, Grover S, Barak T, Shulman LN, Lockman S, Dryden-Peterson S. A Step Toward Timely Referral and Early Diagnosis of Cancer: Implementation and Impact on Knowledge of a Primary Care-Based Training Program in Botswana. Front Oncol. 2018 May 29;8:187. doi: 10.3389/fonc.2018.00187. eCollection 2018. PMID 29896450